CLINICAL TRIAL: NCT00092690
Title: A Multicenter, Double-Blind, Randomized, Parallel Group, 6-Week Study to Evaluate the Efficacy and Safety of Ezetimibe/Simvastatin Combination Tablet Versus Atorvastatin in Patients With Hypercholesterolemia
Brief Title: MK0653A (Ezetimibe (+) Simvastatin) Compared to an Approved Drug (Atorvastatin) for the Treatment of High Cholesterol (0653A-051)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-051; 2004_051
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653A, ezetimibe (+) simvastatin
Drug: Comparator: atorvastatin

SUMMARY:
This study is to assess the safety and efficacy of an investigational drug as compared to an approved drug to reduce specific cholesterol levels.

DETAILED DESCRIPTION:
The duration of treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Elevated cholesterol

Exclusion Criteria:

* Unstable medical conditions or significant heart problems within 3 months prior to first study visit.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1902 (Actual)
Dates: Start 2003-06; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Plasma LDL-C averaged across all doses after 6 weeks

SECONDARY OUTCOMES:
Plasma LDL-C for each dose; plasma HDL-C averaged across all doses

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballantyne CM, Abate N, Yuan Z, King TR, Palmisano J. Dose-comparison study of the combination of ezetimibe and simvastatin (Vytorin) versus atorvastatin in patients with hypercholesterolemia: the Vytorin Versus Atorvastatin (VYVA) study. Am Heart J. 2005 Mar;149(3):464-73. doi: 10.1016/j.ahj.2004.11.023. PMID 15864235
- [Background] Pearson T, Ballantyne C, Sisk C, Shah A, Veltri E, Maccubbin D. Comparison of effects of ezetimibe/simvastatin versus simvastatin versus atorvastatin in reducing C-reactive protein and low-density lipoprotein cholesterol levels. Am J Cardiol. 2007 Jun 15;99(12):1706-1713. doi: 10.1016/j.amjcard.2007.01.062. Epub 2007 May 2. PMID 17560879